CLINICAL TRIAL: NCT00925639
Title: Effects of the Concentrated Extract of Soy on Coagulation Factors After Menopause
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Regiane Helena Barros Rabelo, Departamento de Ginecologia da Universidade Federal de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP/UNIFESP 0728/08
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2009-06-22 (Estimated); Status verified 2009-06

CONDITIONS: Menopause
Keywords: phytoestrogen; coagulation; menopause; ddimer; antithrombin; hypercoagulation
MeSH Terms: conditions — Thrombosis; Thrombophilia | interventions — Isoflavones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isoflavone (Experimental): Patients will receive daily doses of 150 mg of concentrated extract of soy per os
  Interventions: Drug: Isoflavone
- Control (Placebo Comparator): Patients will receive daily placebo pills
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Isoflavone — 150 mg of concentrated extract of soy containing 60 mg of isoflavone comprising 40 mg of genistein, 14,55 mg of daidizein, 3,02 mg of daidzine, 1,14 mg of glicitine, 0,91 mg genistine and 0,38 mg of glicetein.
  Arms: Isoflavone
Drug: Placebo — Starch pill
  Arms: Control

SUMMARY:
Hypoestrogenism, common in menopause, is responsible for systemic and metabolic changes affecting women's wellness, favoring hot flashes, urogenital atrophy and bone mass loss. Hormone reposition therapy (HRT) with estrogen or estrogen associated to progesterone is administered to minimize these effects. Meanwhile, the beneficial effects of HRT are known, there is still concern about its adverse effects such as thromboembolic and cardiovascular effects, increased risk of breast and endometrial cancer. Thus, there is an increasing interest in the development of phytohormonal HRT. The aim of the investigators' study is to evaluate the effects of concentrated extract of soy on hypercoagulation markers in menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* > 1 year of amenorrhea
* 45 to 65 years old
* without hormone reposition treatment or herbal medications in the 6 months preceding the research

Exclusion Criteria:

* history of thromboembolism
* history of cardiovascular disease
* presence of estrogen dependent neoplasia
* presence of abnormal genital bleeding
* uncontrolled metabolic diseases
* smoking or drinking habits
* use of anticoagulants or acetyl salicylic acid

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-01 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Concentration of serum DDimer | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mauro A Aidar, M.D., PhD., Study Chair — Universidade Federal de São Paulo
Locations (1):
- Ambulatório de Ginecologia Endócrina, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: Universidade Federal de Sao Paulo's web page — http://www.unifesp.br